CLINICAL TRIAL: NCT00231998
Title: A Clinical Study Continued From the Confirmatory Study to Validate the Efficacy and Safety of Pimecrolimus Cream in Pediatric Atopic Dermatitis Patients
Brief Title: Extension Study of Pimecrolimus Cream in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981C1302
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, ASM981, pimecrolimus
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel

SUMMARY:
Pimecrolimus, which is an ascomycin derivative, is an anti-inflammatory non-steroidal agent. In this study, the long-term safety and efficacy of Pimecrolimus cream will be evaluated in Japanese pediatric patients with atopic dermatitis. This study is a 6-month extension study following core study.

THIS STUDY IS NOT ENROLLING PATIENTS IN THE UNITED STATES

ELIGIBILITY:
Inclusion Criteria:

* - Patients who had completed the core study and whose participation in this study was considered appropriate as judged by the investigator
* Patients whose guardians have given written informed consent to participation in this study

Exclusion Criteria:

* - Patients who failed in treatment compliance in the core study
* Patients who had a major violation of the protocol in the core study

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 240
Dates: Start 2004-05; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events (AEs)

SECONDARY OUTCOMES:
Number of flares during 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals Japan
Locations (1):
- This study is not being conducted in the United States, Various Cities, Japan